CLINICAL TRIAL: NCT04074122
Title: Electromechanical Profiling of Arrhythmogenic Substrates and Triggers in the Long-QT Syndrome
Brief Title: Electromechanical Profiling of the Long-QT Syndrome (LQTS)
Acronym: EMLoQ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: University of Freiburg (Other); University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 70856
Record Dates: First submitted 2019-07-05; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Long QT Syndrome; Sudden Cardiac Death; Ventricular Tachycardia
Keywords: Electromechanical Mapping; Risk Stratification
MeSH Terms: conditions — Long QT Syndrome; Death, Sudden, Cardiac; Tachycardia, Ventricular | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Symptomatic LQTS patients: Pharmacological (adenosine, epinephrine, isoprenaline) provocation, ECG-imaging and tissue-phase mapping using magnetic resonance imaging (TPM-MRI).
  Interventions: Diagnostic Test: Adenosine and epinephrine, isoprenaline provocation
- Asymptomatic LQTS patients: Pharmacological (adenosine, epinephrine, isoprenaline) provocation, ECG-imaging and tissue-phase mapping using magnetic resonance imaging (TPM-MRI).
  Interventions: Diagnostic Test: Adenosine and epinephrine, isoprenaline provocation
- Healthy controls: Pharmacological (adenosine, epinephrine, isoprenaline) provocation, ECG-imaging and tissue-phase mapping using magnetic resonance imaging (TPM-MRI).
  Interventions: Diagnostic Test: Adenosine and epinephrine, isoprenaline provocation

INTERVENTIONS:
Diagnostic Test: Adenosine and epinephrine, isoprenaline provocation — High-resolution electromechanical mapping at baseline and after provocative measures.
  Other Names: ECG-imaging; Tissue-phase mapping with MRI.

SUMMARY:
High-resolution, non-invasive electromechanical mapping in genotyped long-QT syndrome patients and healthy controls at baseline and during smart provocation.

DETAILED DESCRIPTION:
Using simultaneous ECG-imaging, speckle-tracking analysis and tissue-phase mapping with MRI we will assess electromechanical dispersion at rest. Regional electromechanical elasticity will be investigated during adenosine and epinephrine, isoprenaline infusions and is postulated to increase sudden cardiac death risk prediction in the individual patient.

ELIGIBILITY:
Inclusion Criteria:

LQTS group (Group 1):

* Diagnosis of LQTS according to the ESC guidelines.
* Genetic testing either already performed or consent to genetic testing (at least 5 major LQTS-related genes tested: KCNQ1, KCNH2, SCN5A, KCNE1, KCNE2).

Control group (Group 2):

> Control subjects with structurally normal hearts.

Exclusion Criteria:

* Pregnancy, nursing or planning to become pregnant.
* Known allergy or strong reaction to skin electrodes or contrast agent.
* Inability to give informed consent.
* Presence of metal objects in or attached to the body.
* Dialysis.
* Cardiomyopathy.
* Second-degree heart block or higher degrees of block.
* Sick sinus syndrome.
* Asthma.
* Chronic obstructive pulmonary disease.
* Left-main coronary artery disease.
* Unstable coronary artery disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation.
Study Population: Potential study subjects will be selected from the Cardiogenetic or Cardiac Outpatient Clinic or during their in-hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Differences in regional electromechanical dispersion between LQTS patients and controls | At day of investigation
  Electromechanical dispersion in milliseconds
Differences in regional electromechanical dispersion between symptomatic and asymptomatic LQTS patients | At day of investigation
  Electromechanical dispersion in milliseconds

SECONDARY OUTCOMES:
Correlation of electromechanical dispersion between LQTS type 1, 2, and 3. | At day of investigation
  Electromechanical dispersion in milliseconds
Relation between global electromechanical window vs regional electromechanical dispersion in LQTS | At day of investigation
  Electromechanical dispersion in milliseconds
Correlation between mechanical dispersion using TPM-MRI and cine-MRI | At day of investigation
  Time-to-diastolic peak in milliseconds
Correlation between mechanical dispersion using TPM-MRI and speckle-tracking echocardiography | At day of investigation
  Time-to-peak in milliseconds

CONTACTS AND LOCATIONS:
Overall Officials: Paul Volders, MD, PhD, Principal Investigator — Maastricht UMC

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Haugaa KH, Edvardsen T, Leren TP, Gran JM, Smiseth OA, Amlie JP. Left ventricular mechanical dispersion by tissue Doppler imaging: a novel approach for identifying high-risk individuals with long QT syndrome. Eur Heart J. 2009 Feb;30(3):330-7. doi: 10.1093/eurheartj/ehn466. Epub 2008 Oct 21. PMID 18940888
- [Result] Haugaa KH, Amlie JP, Berge KE, Leren TP, Smiseth OA, Edvardsen T. Transmural differences in myocardial contraction in long-QT syndrome: mechanical consequences of ion channel dysfunction. Circulation. 2010 Oct 5;122(14):1355-63. doi: 10.1161/CIRCULATIONAHA.110.960377. Epub 2010 Sep 20. PMID 20855658
- [Result] ter Bekke RM, Volders PG. Arrhythmogenic mechano-electric heterogeneity in the long-QT syndrome. Prog Biophys Mol Biol. 2012 Oct-Nov;110(2-3):347-58. doi: 10.1016/j.pbiomolbio.2012.07.007. Epub 2012 Jul 24. PMID 22841828
- [Result] ter Bekke RM, Haugaa KH, van den Wijngaard A, Bos JM, Ackerman MJ, Edvardsen T, Volders PG. Electromechanical window negativity in genotyped long-QT syndrome patients: relation to arrhythmia risk. Eur Heart J. 2015 Jan 14;36(3):179-86. doi: 10.1093/eurheartj/ehu370. Epub 2014 Sep 8. PMID 25205533
- [Result] Shimizu W, Antzelevitch C. Differential effects of beta-adrenergic agonists and antagonists in LQT1, LQT2 and LQT3 models of the long QT syndrome. J Am Coll Cardiol. 2000 Mar 1;35(3):778-86. doi: 10.1016/s0735-1097(99)00582-3. PMID 10716483
- [Result] Viskin S, Rosso R, Rogowski O, Belhassen B, Levitas A, Wagshal A, Katz A, Fourey D, Zeltser D, Oliva A, Pollevick GD, Antzelevitch C, Rozovski U. Provocation of sudden heart rate oscillation with adenosine exposes abnormal QT responses in patients with long QT syndrome: a bedside test for diagnosing long QT syndrome. Eur Heart J. 2006 Feb;27(4):469-75. doi: 10.1093/eurheartj/ehi460. Epub 2005 Aug 16. PMID 16105845